CLINICAL TRIAL: NCT03023657
Title: Detection of Arousal With Facial Micro-expression in Severe Brain-damaged Patient
Acronym: DAME
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties to realize the protocol
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1608177; 2016-A01973-48 (Other: ANSM)
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Consciousness Disorder
Keywords: arousal; Consciousness Disorders; vegetative state; minimally conscious state
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe brain-damaged patient in coma awakening (Experimental): For each patient, video sessions of the face will be performed during a waking period, until the spontaneous macro-EFE (Emotional Facial Expression) reappears. The video sessions will be done without stimulation or with visual, auditory or tactile stimulation. The sessions will be daily for 7 days then weekly for a maximum duration of 4 weeks.
  Interventions: Other: Detection of arousal

INTERVENTIONS:
Other: Detection of arousal — Detecting facial microexpression before visible facial expressions in patient with disorder of consciousness after severe brain injury

SUMMARY:
Severe brain injuries lead to disorders of consciousness after coma. During this awakening period, detection of arousal is critical to the adaptation of medical strategy, but global paralysis, including facial expression, make the clinical assessment very difficult. Emotional facial expressions are a significant part of this clinical assessment. They are both a landmark of the internal state of the patient (comfort versus discomfort) and a landmark of the relational level with his environment. Visible emotional facial expression is a large temporal phenomenon lasting a couple of seconds, while a microexpression is barely noticeable and very brief. These micro expressions are usually produced when one tried to voluntary hide emotional expressions. In this study, we hypothesize that some patients awakening from coma could still produce microexpression before being able to produce visible emotional facial expressions. This ability to produce micro-expression could be an early landmark of relational awakening in severe brain lesions.

ELIGIBILITY:
Inclusion Criteria:

* Brain-damaged patient (stroke, traumatic brain injury, anoxia)
* Disorder of consciousness (CRS-R≤ 10) more than 48h after stopping sedation
* Patient without spontaneous or stimulated facial expressions

Exclusion Criteria:

* Medically unstable patient

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
facial micro expression found in at least one patient on one video recording | Every day for a week then once a week for four weeks
  Optical camera and thermal camera

CONTACTS AND LOCATIONS:
Overall Officials: Pascal GIRAUX, MDPhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - Chu Saint-Etienne, Saint-Etienne
  - Clinique Mutualiste Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No